CLINICAL TRIAL: NCT06539650
Title: Neural Adaptations to a Single Session Metronome-Paced Strength Training: Insights From Neuroscience and Human Movement Variability
Brief Title: Neural Adaptations to a Single Session of Metronome-Paced Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); University of Essex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AcuteMETROTRAIN - 1404
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Motor Control; Neuroscience; Neural Adapatations; Transcranial Magnetic Stimulation; Dynamic Systems; Metronome Paced Strength Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractal Paced (Experimental): Strength training in single leg extension machine, synchronizing each repetition with a fractal-like visual metronome, i.e., a metronome presenting visual external cues with variability within its temporal structure.
  Interventions: Other: Fractal Paced
- Isochronous Paced (Experimental): Strength training in single leg extension machine, synchronizing each repetition with a isochronus visual metronome, i.e., a metronome presenting visual external cues withthe same pace in each repetition (without variability)
  Interventions: Other: Isochronus Paced
- Self Paced (Experimental): Strength training in single leg extension machine at participants self pace.
  Interventions: Other: Self Paced

INTERVENTIONS:
Other: Fractal Paced — The intervention consists in a single session of metronome paced strength training composed by 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) in single leg extension machine, synchronizing each repetition with fractal external cues presented by a visual metronome. The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Fractal Paced
Other: Isochronus Paced — The intervention consists in a single session of metronome paced strength training composed by 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) in single leg extension machine, synchronizing each repetition with isochronus external cues presented by a visual metronome. The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Isochronous Paced
Other: Self Paced — The intervention consists in a single session of strength training composed by 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) in single leg extension machine, at at participants' own self pace (with no metronome). The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Self Paced

SUMMARY:
The aim of the study is to investigate the effects of incorporating variability within a single session of Resistance Training (RT) methods on the neural adaptations along the corticospinal tract and on neuromuscular function. The literature suggests that RTis one of the most common modalities to enhance and restore muscle function and its practice results in adaptation in neural and morphological adaptations. Moreover, it is also known that muscle contraction relies on the coordination and regulation of the descending neural drive from the motor cortex to the motoneurons and from the motoneurons to the muscles. However, traditional RT programs tend not to address this motor control dimension. Recent approaches such as metronome paced strength training have been used to cover this motor control dimension through a greater control and consciousness of movement. However, this methodology tends not to incorporate the inherent variability and complex, fractal-like fluctuations that characterize human movement. The investigators propose that incorporating variability through a fractal-like metronome approach will speed up the neural adaptations which will be useful in injury rehab

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* aged between 18 and 40 years

Exclusion Criteria:

* Neurologic conditions;
* Lower limb disabilities or disease;
* Not able to provide informed consent;
* Have an implanted device (e.g. pacemakers) or any metal in the body;
* Medication advised against the application of Transcranial Magnetic Stimulation;
* History/family history of seizures, brain lesions or head trauma, neurological or psychiatric diseases, epilepsy, migraine

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Corticospinal Excitability (CSE) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  CSE is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of excitability of the corticospinal tract.
Short-Interval Intracortical Inhibition (SICI) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  SICI is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of inhibition within the motor cortex.
Corticospinal Silent Period (CSP) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  CSP is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of inhibition along the corticospinal tract.
Intracortical Facilitation (ICF) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  ICF is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of facilitation within the motor cortex.
Lumbar Evoked Potentials (LEP) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  LEP is a measure extracted through the aplication of Lumbar stimulation. This measure allow to distinguish the adaptations that occur at spinal level as a result of strength training.
Maximal Compound Action Potentials (Mmax) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  Mmax is a measure assessed through peripheral nerve stimulation and represents the maximal capacity of recruit the motoneurons that innerve a muscle

SECONDARY OUTCOMES:
Maximal Voluntary Isometric Contraction (MVIC) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  MVIC is defined as the maximal force an individual can produce against an immovable resistance
Sample Entropy (SampEn) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  SampEn is a non-linear measure of the temporal structure of force output, being an indicator of the regularity of this physiological output. It is obtained from sustained submaximal isometric contractions and it has been proposed as an indirect index of the capacity of the neuromuscular system to adapt the force output to changes in environment, i.e., its adaptability.
Coefficient ov variation (CV) changes Pre-to-Post intervention both within and between Fractal paced, Isochronus Paced and Self paced conditions | PRE (before intervention), POST (immediately after the intervention) and POST 60 (60 minutes after the intervention)
  CV is a common linear measure that translates the amount of variability within the signal and is calculated through the standard deviation normalised to the mean of a time series

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health & Science, Almada, Monte de Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No